CLINICAL TRIAL: NCT01554137
Title: Interests of Strengthening Isokinetic Upper Extremity Hemiparetic Sequelae in Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 8571
Record Dates: First submitted 2012-03-12; First posted 2012-03-14 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Partial Deficiency of Muscle Strength
MeSH Terms: interventions — Range of Motion, Articular

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- With isokinetic strength training (Experimental): 60 minutes isokinetic strength training on concentric mode
  Interventions: Other: isokinetic strength training
- without isokinetic strength training (Placebo Comparator): passive motion 60 minutes
  Interventions: Other: passive motion

INTERVENTIONS:
Other: isokinetic strength training — The experimental group will follow a program of 18 sessions (3 sessions per week for 6 weeks) with a physiotherapy treatment (30 minutes) and occupational therapy (30 minutes), and a building session isokinetic concentric mode extensor and flexor muscles of the elbow extensors and wrist flexors.
  Arms: With isokinetic strength training
Other: passive motion — The control group will follow a program of 18 sessions of physiotherapy and occupational therapy combined with 18 sessions of passive motion in flexion-elbow extension, wrist flexion-extension on the isokinetic device
  Arms: without isokinetic strength training

SUMMARY:
Stroke (CVA) is the leading cause of death and the leading cause of disability in developed countries as in developing countries (WHO, 2000). In the aftermath of a stroke, patients keep a permanent disability in 75% of cases and only one quarter of them is able to resume work. The post stroke sequelae are sensory-motor and cognitive.

According to literature data, 75-83% of patients who survive a stroke learn to walk only 25 to 45% recover use of their upper limb in activities of daily living (Friedman, 1990).

The existence of a phase called "plateau" in motor recovery after stroke has been suggested (Colautti, 2001). This would occur beyond the 4 th month and would correspond to a phase where the rehabilitation techniques used in the subacute phase are deemed less effective. Recently, Page (2004) speculated that this plateau phase is rather the consequence of adaptation to the type of patient follow-up training and not that of a limit to the possibilities of recovery. In an observational study on the recovery of upper limb conducted over a period of 4 years, Broeks (2004) showed a possible recovery beyond 16 weeks post stroke. The results of studies on different techniques for rehabilitation of chronic stroke patients tend to confirm the hypothesis of page. Therefore, varying the training parameters (type, intensity, frequency) could improve the functional capabilities of these patients, even at a distance of stroke.

Strength training is part of the management of hemiparetic patients. The results of several studies show an improvement in muscle strength and functional ability to walk after a building program isokinetic lower limb (Sharp, 1997).

The objective of our project is to evaluate the effectiveness of a building program of isokinetic muscle on the paretic limb motor recovery in hemiparetic patients over 6 months of a stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patients with more than 6 months post stroke,
* Muscular control greater than or equal to 3 on the extensors and elbow flexors,
* Muscular control greater than or equal to 3 on the flexors and extensors of the wrist,
* Spasticity less than or equal to 3 on the muscle groups mentioned above, s
* Active abduction of the shoulder above 60 ° and painless
* Absence of cognitive impairment (MMS> 22 without any trouble phasic)
* No orthopedic limitations at the elbow and wrist,

Exclusion Criteria:

* Progressive neurological or systemic involvement,
* Orthopedic limitations at the elbow or wrist
* Cognitive,
* Hemineglect,
* Severe aphasia with impaired comprehension,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
upper limb motor function | 6 weeks
  improving upper limb motor recovery at the end of the program is evaluated by the Fugl-Meyer test.This test evaluates motor impairment of the hemiplegic upper limb, balance, sensitivity, passive joint mobility and joint pain at mobilization.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia COROIAN, MD, Principal Investigator — UH Montpellier
Locations (1):
- Service de médecine Physique et de Réadaptation, Montpellier, France

REFERENCES:
- [Derived] Coroian F, Jourdan C, Bakhti K, Palayer C, Jaussent A, Picot MC, Mottet D, Julia M, Bonnin HY, Laffont I. Upper Limb Isokinetic Strengthening Versus Passive Mobilization in Patients With Chronic Stroke: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2018 Feb;99(2):321-328. doi: 10.1016/j.apmr.2017.08.490. Epub 2017 Sep 22. PMID 28947166